

## **Consent to Participate in Research**

## A study on social event, mental health and family relationship

| I hereby cor | nsent to participate in the captioned research con | ducted by Di |
|---|---|---|
| Herman Lo, Associate Professor, Polytechnic University. | Department of Applied Social Sciences, The | Hong Kong |
| | ned from this research may be used in future rivacy will be retained, i.e. my personal details | |
| * | thed information sheet has been fully explained. articipation in the project is voluntary. | I understand |
| I acknowledge that I have the right t time without penalty of any kind. | o question any part of the procedure and can wit | hdraw at any |
| Name of Participant | | |
| Signature of Participant | | |
| Name of Principal Investigator | 盧希皿博士 | |
| Signature of Principal Investigator | | |
| Date | | |